CLINICAL TRIAL: NCT01243944
Title: Randomized, Open Label, Multicenter Phase III Study of Efficacy and Safety in Polycythemia Vera Subjects Who Are Resistant to or Intolerant of Hydroxyurea: JAK Inhibitor INC424 Tablets Versus Best Available Care (The RESPONSE Trial)
Brief Title: Study of Efficacy and Safety in Polycythemia Vera Subjects Who Are Resistant to or Intolerant of Hydroxyurea: JAK Inhibitor INC424 (INCB018424) Tablets Versus Best Available Care: (The RESPONSE Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC424B2301
Expanded Access: NCT03147742 (Approved for marketing)
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Polycythemia Vera
Keywords: INCB018424
MeSH Terms: conditions — Polycythemia Vera | interventions — ruxolitinib; Hydroxyurea; Pipobroman; anagrelide; Lenalidomide; pomalidomide

ARMS (2):
- ruxolitinib tablets (Experimental): Starting dose of 10 mg BID with individualized dose titration ranging from 5 mg once a day (QD) to 25 mg BID based on safety and efficacy
  Interventions: Drug: ruxolitinib tablets
- Best Available Therapy (Other): Best Available Therapy (BAT) will be selected by the Investigator for each participant. BAT may not include experimental agents (i.e. those not approved for the treatment of any indication) as well as a limited number of other selected drugs in accordance with the protocol-defined requirements.
  Interventions: Other: Best Available Therapy (BAT)

INTERVENTIONS:
Drug: ruxolitinib tablets — Starting dose of 10 mg BID with individualized dose titration ranging from 5 mg QD to 25 mg BID based on safety and efficacy
  Arms: ruxolitinib tablets
Other: Best Available Therapy (BAT) — Best Available Therapy (BAT) will be selected by the Investigator for each participant. BAT may not include experimental agents (i.e. those not approved for the treatment of any indication) as well as a limited number of other selected drugs in accordance with the protocol-defined requirements.
  Other Names: BAT could include:; Hydroxyurea; IFN/PEG-IFN; Pipobroman; Anagrelide; Lenalidomide; Pomalidomide; Observation only
  Arms: Best Available Therapy

SUMMARY:
This pivotal phase III trial (CINC424B2301) is designed to compare the efficacy and safety of ruxolitinib (INC424) to Best Available Therapy (BAT) in participants with polycythemia vera (PV) who are resistant to or intolerant of hydroxyurea (HU).

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with PV for at least 24 weeks prior to screening according to the 2008 World Health Organization criteria
* Participants resistant to or intolerant of hydroxyurea
* Participants with a phlebotomy requirement
* Participants with splenomegaly (palpable or non-palpable) and a spleen volume, as measured by MRI (or CT in applicable participants ), of greater than or equal to 450 cubic centimeters
* Participants with an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2

Exclusion Criteria:

* Women who are pregnant or nursing
* Participants with inadequate liver or renal function
* Participants with significant bacterial, fungal, parasitic, or viral infection requiring treatment
* Participants with an active malignancy within the past 5 years, excluding specific skin cancers
* Participants with known active hepatitis or HIV positivity
* Participants who have previously received treatment with a JAK inhibitor
* Participants being treated with any investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2010-10-27 (Actual); Primary Completion 2014-01-15 (Actual); Study Completion 2018-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, MD,PhD, Study Director — M.D. Anderson Cancer Center; Mark Jones, MD, Study Director — Incyte Corporation
Locations (102):
- United States (28):
  - Birmingham, Alabama
  - Scottsdale, Arizona
  - Pomona, California
  - Sacramento, California
  - San Diego, California
  - Bridgeport, Connecticut
  - New Haven, Connecticut
  - Boynton Beach, Florida
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Winter Park, Florida
  - Boise, Idaho
  - Chicago, Illinois
  - Lafayette, Louisiana
  - Scarborough, Maine
  - Baltimore, Maryland
  - Columbia, Maryland
  - Southfield, Michigan
  - Jefferson City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Morristown, New Jersey
  - Somerville, New Jersey
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - Seattle, Washington
- Buenos Aires, Argentina
- Australia (3):
  - Brisbane
  - Parkville
  - Tweed Heads
- Belgium (4):
  - Antwerp
  - Bruges
  - Brussels
  - Leuven
- Canada (3):
  - Hamilton
  - Montreal
  - Toronto
- China (2):
  - Beijing
  - Hangzhou
- France (7):
  - Avignon
  - Bayonne
  - Brest
  - Lille
  - Nantes
  - Paris
  - Vandœuvre-lès-Nancy
- Germany (11):
  - Aachen
  - Berlin
  - Bonn
  - Freiburg im Breisgau
  - Hamburg
  - Jena
  - Magdeburg
  - Mannheim
  - Minden
  - München
  - Ulm
- Hungary (4):
  - Budapest
  - Kecskemét
  - Szeged
  - Szombathely
- Italy (12):
  - Bari
  - Bergamo
  - Bologna
  - Florence
  - Milan
  - Napoli
  - Orbassano
  - Pavia
  - Reggio Calabria
  - Roma
  - Varese
  - Vicenza
- Japan (6):
  - Chiba
  - Chuo-city Yamanashi
  - Maebashi
  - Nagoya-city Aichi
  - Osaka
  - Tokyo
- Netherlands (2):
  - Enschede
  - Rotterdam
- Russia (2):
  - Moscow
  - Saint Petersburg
- Seoul, South Korea
- Spain (9):
  - A Coruña
  - Barcelona
  - Las Palmas de Gran Canaria
  - Madrid
  - Majadahonda
  - Málaga
  - Pamplona
  - Salamanca
  - Valencia
- Bangkok, Thailand
- Turkey (Türkiye) (3):
  - Ankara
  - Istanbul
  - Izmir
- United Kingdom (3):
  - Bournemouth
  - Cardiff
  - London

REFERENCES:
- [Derived] Kiladjian JJ, Zachee P, Hino M, Pane F, Masszi T, Harrison CN, Mesa R, Miller CB, Passamonti F, Durrant S, Griesshammer M, Kirito K, Besses C, Moiraghi B, Rumi E, Rosti V, Blau IW, Francillard N, Dong T, Wroclawska M, Vannucchi AM, Verstovsek S. Long-term efficacy and safety of ruxolitinib versus best available therapy in polycythaemia vera (RESPONSE): 5-year follow up of a phase 3 study. Lancet Haematol. 2020 Mar;7(3):e226-e237. doi: 10.1016/S2352-3026(19)30207-8. Epub 2020 Jan 23. PMID 31982039
- [Derived] Kiladjian JJ, Guglielmelli P, Griesshammer M, Saydam G, Masszi T, Durrant S, Passamonti F, Jones M, Zhen H, Li J, Gadbaw B, Perez Ronco J, Khan M, Verstovsek S. Efficacy and safety of ruxolitinib after and versus interferon use in the RESPONSE studies. Ann Hematol. 2018 Apr;97(4):617-627. doi: 10.1007/s00277-017-3225-1. Epub 2018 Feb 2. PMID 29396713
- [Derived] Verstovsek S, Harrison CN, Kiladjian JJ, Miller C, Naim AB, Paranagama DC, Habr D, Vannucchi AM. Markers of iron deficiency in patients with polycythemia vera receiving ruxolitinib or best available therapy. Leuk Res. 2017 May;56:52-59. doi: 10.1016/j.leukres.2017.01.032. Epub 2017 Jan 31. PMID 28193568
- [Derived] Verstovsek S, Vannucchi AM, Griesshammer M, Masszi T, Durrant S, Passamonti F, Harrison CN, Pane F, Zachee P, Kirito K, Besses C, Hino M, Moiraghi B, Miller CB, Cazzola M, Rosti V, Blau I, Mesa R, Jones MM, Zhen H, Li J, Francillard N, Habr D, Kiladjian JJ. Ruxolitinib versus best available therapy in patients with polycythemia vera: 80-week follow-up from the RESPONSE trial. Haematologica. 2016 Jul;101(7):821-9. doi: 10.3324/haematol.2016.143644. Epub 2016 Apr 21. PMID 27102499
- [Derived] Vannucchi AM, Kiladjian JJ, Griesshammer M, Masszi T, Durrant S, Passamonti F, Harrison CN, Pane F, Zachee P, Mesa R, He S, Jones MM, Garrett W, Li J, Pirron U, Habr D, Verstovsek S. Ruxolitinib versus standard therapy for the treatment of polycythemia vera. N Engl J Med. 2015 Jan 29;372(5):426-35. doi: 10.1056/NEJMoa1409002. PMID 25629741

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants may be treated beyond 256 weeks due to the 14 day visit window.
Groups:
- Ruxolitinib: Starting dose of 10 mg twice a day (BID) with individualized dose titration ranging from 5 mg once a day (QD) to 25 mg BID based on safety and efficacy
Period: Overall Study
Arm/Group | Ruxolitinib | Best Available Therapy
Started | 110 | 112 (One participant withdrew consent 5 days after randomization to BAT & wasn't treated while on study.)
Treated | 110 | 111
Followed for Survival | 22 | 21
Completed | 65 | 61 (Study evaluation completion is reported for participants that were treated & those never treatment.)
Not Completed | 45 | 51
Not completed — Adverse Event | 15 | 13
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 2 | 7
Not completed — Disease progression | 12 | 11
Not completed — Protocol deviation | 1 | 1
Not completed — Participant decision | 10 | 15
Not completed — Death | 2 | 3
Not completed — Non-compliance with study treatment | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants, regardless treated or not.
Groups:
- Ruxolitinib: Starting dose of 10 mg BID with individualized dose titration ranging from 5 mg QD to 25 mg BID based on safety and efficacy
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib | Best Available Therapy | Total
Number analyzed (Participants) | 110 | 112 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (10.48) | 59.1 (10.25) | 60.1 (10.39)
Age, Customized [Number; unit: participants]
  < 60 years | 49 | 54 | 103
  ≥ 60 years | 61 | 58 | 119
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 32 | 76
  Male | 66 | 80 | 146
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 98 | 96 | 194
  Black/African American | 1 | 0 | 1
  Asian | 11 | 16 | 27
Weight [Mean (Standard Deviation); unit: kg] | 76.6 (14.09) | 79.0 (17.34) | 77.8 (15.83)
Height [Mean (Standard Deviation); unit: cm] — Height was missing at study entry for one participant in the ruxolitinib arm.
  cm | 172.2 (8.44) | 173.3 (9.79) | 172.8 (9.14)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.8 (3.82) | 26.1 (4.24) | 25.9 (4.03)
ECOG performance status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) - ECOG Status: 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=Ambulatory and capable of all selfcare but unable to carry out any work activities up and about more than 50% of waking hours
  participants
    0 | 76 | 77 | 153
    1 | 31 | 34 | 65
    2 | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Achieving a Primary Response at Week 32
Description: Primary response was defined as having achieved hematocrit control (the absence of phlebotomy eligibility beginning at the Week 8 visit and continuing through Week 32) and Spleen Volume Reduction (a greater than or equal to 35% reduction from baseline in spleen volume at Week 32).
Time Frame: 32 Weeks
Population: Full Analysis Set (FAS) comprises all participants to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 110 | 112
percentage of participants | 22.7 [15.3 to 31.7] | 0.9 [0.0 to 4.9]
Statistical Analysis 1: Comparison: Ruxolitinib vs Best Available Therapy; Test type: Superiority or Other; p < 0.0001, Exact Cochran-Mantel-Haenszel; Odds Ratio, log = 32.67, 95% CI 2-sided [5.04 to 1337]

2. Secondary Outcome: The Percentage of Participants Achieving a Durable Primary Response at Week 48
Description: Durable Primary Response was defined as any participant who achieved the primary outcome measure and who maintained their response up to 48 weeks after randomization.
Time Frame: 48 Weeks
Population: Full Analysis Set (FAS) comprises all participants to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 110 | 112
percentage of participants | 20.0 [13.0 to 28.7] | 0.9 [0.0 to 4.9]
Statistical Analysis 1: Comparison: Ruxolitinib vs Best Available Therapy; Test type: Superiority or Other; p < 0.0001, Exact Cochran-Mantel-Haenszel; Odds Ratio (OR) = 28.01, 95% CI 2-sided [4.24 to 1144]

3. Secondary Outcome: The Percentage of Participants Achieving Complete Hematological Remission at Week 32
Description: Complete Hematological Remission at Week 32 was defined as any participant who achieved hematocrit control with a platelet count less than or equal to 400 X 10^9/L and a white blood cell count less than or equal to 10 X 10^9/L.
Time Frame: 32 Weeks
Population: Full Analysis Set (FAS) comprises all participants to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 110 | 112
percentage of participants | 23.6 [16.1 to 32.7] | 8.0 [3.7 to 14.7]
Statistical Analysis 1: Comparison: Ruxolitinib vs Best Available Therapy; Test type: Superiority or Other; p = 0.0016, Exact Cochran-Mantel-Haenszel; P-value was calculated using stratified exact Cochran-Mantel-Haenszel test by adjusting for the WBC/platelet status (abnormal vs normal) at baseline; Odds Ratio (OR) = 3.57, 95% CI 2-sided [1.50 to 9.06]

4. Secondary Outcome: The Percentage of Participants Who Achieved a Durable Complete Hematological Remission at Week 48
Description: Durable Complete Hematological Remission was defined as any participant who achieved Complete Hematological Remission at Week 32 and maintained their response up to 48 weeks after randomization.
Time Frame: 48 Weeks
Population: Full Analysis Set (FAS) comprises all participants to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 110 | 112
percentage of participants | 20.9 [13.7 to 29.7] | 0.9 [0.0 to 4.9]

5. Secondary Outcome: The Percentage of Participants Who Achieved a Durable Hematocrit Control at Week 48
Description: Durable Hematocrit Control was defined as any participant who achieved phlebotomy eligibility independence from Week 8 to Week 32 and maintained hematocrit control up to 48 weeks after randomization.
Time Frame: 48 Weeks
Population: Full Analysis Set (FAS) comprises all participants to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 110 | 112
percentage of participants | 54.5 [44.8 to 64.1] | 1.8 [0.2 to 6.3]

6. Secondary Outcome: The Percentage of Participants Who Achieved Durable Spleen Volume Reduction at Week 48
Description: Durable Spleen Volume Reduction was defined as a participant who achieved at least 35% reduction from baseline in spleen volume at Week 32 and maintained that response 48 weeks after randomization.
Time Frame: 48 Weeks
Population: Full Analysis Set (FAS) comprises all participants to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 110 | 112
percentage of participants | 37.3 [28.2 to 47.0] | 0.9 [0.0 to 4.9]

7. Secondary Outcome: Estimated Duration of the Primary Response
Description: Duration of the primary response is defined as the time from the first occurrence when both components of the primary endpoint are met until the date of the first documented disease progression (end of response).
  Kaplan-Meier estimates are provided for duration of primary response.
Time Frame: Through study completion, analysis was conducted when all participants had completed the Week 80 visit or discontinued the study
Population: Full Analysis Set (FAS) comprises all participants to whom study treatment had been assigned by randomization. Duration of response was pre-specified in the protocol to be analyzed for the ruxolitinib arm only considering the study design which allowed crossover for the BAT arm beginning at Week 32.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 110
probability
  16 weeks | 1.00 [NA to NA] — A confidence interval cannot be estimated at this time-point because no one had lost response.
  32 weeks | 1.00 [NA to NA] — A confidence interval cannot be estimated at this time-point because no one had lost response.
  48 weeks | 0.92 [0.72 to 0.98]
  64 weeks | 0.92 [0.72 to 0.98]
  80 weeks | 0.92 [0.72 to 0.98]
  96 weeks | 0.88 [0.67 to 0.96]
  112 weeks | 0.84 [0.62 to 0.94]
  128 weeks | 0.84 [0.62 to 0.94]
  144 weeks | 0.84 [0.62 to 0.94]
  160 weeks | 0.79 [0.57 to 0.91]
  176 weeks | 0.79 [0.57 to 0.91]
  192 weeks | 0.74 [0.51 to 0.88]
  208 weeks | 0.74 [0.51 to 0.88]
  224 weeks | 0.74 [0.51 to 0.88]
  240 weeks | NA [NA to NA] — No additional progression was experienced within population at week 240.
  256 weeks | NA [NA to NA] — No additional progression was experienced within population at week 256.

8. Secondary Outcome: The Percentage of Participants Who Achieved Overall Clinicohematologic Response at Week 32
Description: Overall Clinicohematologic Response is defined as any participant who achieved a complete or partial clinicohematologic response per the European LeukemiaNet modified criteria for response in polycythemia vera (PV). A Complete Response (CR) is defined as: hematocrit control, spleen volume reduction at least 35% from baseline, platelet count less than or equal to 400 x 10(9)/L, and white blood cell count less than or equal to 10 x 10(9)/L. A Partial Response (PR) is defined as hematocrit control or response in all 3 of the other criteria.
Time Frame: 32 Weeks
Population: Full Analysis Set (FAS) comprises all participants to whom study treatment had been assigned by randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 110 | 112
percentage of participants
  Complete response rate | 8.2 | 0.9
  Partial response rate | 54.5 | 18.8

9. Secondary Outcome: The Percentage of Participants Achieving a Durable Complete or Partial Clinicohematologic Response at Week 48
Description: Durable Complete or Partial Clinicohematologic Response was defined as any participant who achieved complete or partial clinicohematologic response per the European LeukemiaNet modified criteria for response in polycythemia vera at Week 32 and maintained that response 48 weeks after randomization.
Time Frame: 48 Weeks
Population: Full Analysis Set (FAS) comprises all participants to whom study treatment had been assigned by randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 110 | 112
percentage of participants
  Complete response rate | 7.3 | 0.9
  Partial response rate | 50.9 | 0.9

10. Secondary Outcome: Estimated Duration of the Complete Hematological Remission
Description: Duration of the complete hematological remission is defined as the time from the first occurrence of complete hematological remission until the date of the first documented progression (end of response).
  Kaplan-Meier estimates are provided for duration of complete hematological remission.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 110
probability
  16 weeks | 1.00 [NA to NA] — A confidence interval cannot be estimated at this time-point because no one had lost response.
  32 weeks | 1.00 [NA to NA] — A confidence interval cannot be estimated at this time-point because no one had lost response.
  48 weeks | 0.88 [0.66 to 0.96]
  64 weeks | 0.83 [0.61 to 0.93]
  80 weeks | 0.74 [0.51 to 0.87]
  96 weeks | 0.74 [0.51 to 0.87]
  112 weeks | 0.69 [0.46 to 0.84]
  128 weeks | 0.69 [0.46 to 0.84]
  144 weeks | 0.65 [0.41 to 0.81]
  160 weeks | 0.65 [0.41 to 0.81]
  176 weeks | 0.55 [0.32 to 0.73]
  192 weeks | 0.55 [0.32 to 0.73]
  208 weeks | 0.55 [0.32 to 0.73]
  224 weeks | 0.55 [0.32 to 0.73]
  240 weeks | NA [NA to NA] — No additional progression was experienced within population at week 240.
  256 weeks | NA [NA to NA] — No additional progression was experienced within population at week 256.

11. Secondary Outcome: Duration of the Absence of Phlebotomy Eligibility
Description: Duration of the absence of phlebotomy eligibility is defined as the time from the first occurrence of absence of phlebotomy eligibility until the date of the first documented progression.
Time Frame: 256 Weeks
Population: Full Analysis Set (FAS) comprises all participants to whom study treatment had been assigned by randomization. Duration of the absence of phlebotomy eligibility was pre-specified in the protocol to be analyzed for the ruxolitinib arm only considering the study design which allowed crossover for the BAT arm beginning at Week 32.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 110
probability
  16 weeks | 1.00 [NA to NA] — A confidence interval cannot be estimated at this time-point because no one had lost response.
  32 weeks | 1.00 [NA to NA] — A confidence interval cannot be estimated at this time-point because no one had lost response.
  48 weeks | 0.97 [0.88 to 0.99]
  64 weeks | 0.92 [0.82 to 0.97]
  80 weeks | 0.91 [0.80 to 0.96]
  96 weeks | 0.91 [0.80 to 0.96]
  112 weeks | 0.87 [0.76 to 0.93]
  128 weeks | 0.84 [0.72 to 0.91]
  144 weeks | 0.84 [0.72 to 0.91]
  160 weeks | 0.82 [0.70 to 0.90]
  176 weeks | 0.79 [0.66 to 0.87]
  192 weeks | 0.77 [0.64 to 0.86]
  208 weeks | 0.73 [0.60 to 0.83]
  224 weeks | 0.73 [0.60 to 0.83]
  240 weeks | 0.73 [0.60 to 0.83]
  256 weeks | 0.73 [0.60 to 0.83]

12. Secondary Outcome: Duration of Reduction in Spleen Volume
Description: Duration of spleen volume reduction is defined as the time from the first occurrence of a >=35% reduction from baseline in spleen volume until the date of the first documented progression.
Time Frame: 256 Weeks
Population: Full Analysis Set (FAS) comprises all participants to whom study treatment had been assigned by randomization. Duration of the reduction in spleen volume was pre-specified in the protocol to be analyzed for the ruxolitinib arm only considering the study design which allowed crossover for the BAT arm beginning at Week 32.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 110
probability
  16 weeks | 1.00 [NA to NA] — A confidence interval cannot be estimated at this time-point because none of the participants had progressed.
  32 weeks | 1.00 [NA to NA] — A confidence interval cannot be estimated at this time-point because none of the participants had progressed.
  48 weeks | 1.00 [NA to NA] — A confidence interval cannot be estimated at this time-point because none of the participants had progressed.
  64 weeks | 1.00 [NA to NA] — A confidence interval cannot be estimated at this time-point because none of the participants had progressed.
  80 weeks | 1.00 [NA to NA] — A confidence interval cannot be estimated at this time-point because none of the participants had progressed.
  96 weeks | 0.98 [0.84 to 1.00]
  112 weeks | 0.95 [0.82 to 0.99]
  128 weeks | 0.95 [0.82 to 0.99]
  144 weeks | 0.95 [0.82 to 0.99]
  160 weeks | 0.93 [0.79 to 0.98]
  176 weeks | 0.93 [0.79 to 0.98]
  192 weeks | 0.93 [0.79 to 0.98]
  208 weeks | 0.87 [0.66 to 0.95]
  224 weeks | 0.72 [0.34 to 0.91]
  240 weeks | NA [NA to NA] — No additional progression was experienced within population at week 240.
  256 weeks | NA [NA to NA] — No additional progression was experienced within population at week 256.

13. Secondary Outcome: Duration of The Overall Clinicohematologic Response
Description: Duration of the overall clinicohematologic response was defined as the time from the first occurrence of complete response (CR) or partial response (PR) until the date of the first documented disease progression.
Time Frame: 256 Weeks
Population: Full Analysis Set (FAS) comprises all participants to whom study treatment had been assigned by randomization. Duration of the overall clinicohematologic response was pre-specified in the protocol to be analyzed for the ruxolitinib arm only considering the study design which allowed crossover for the BAT arm beginning at Week 32.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 110
probability
  16 weeks | 1.00 [NA to NA] — A confidence interval cannot be estimated at this time-point because no one had lost response.
  32 weeks | 0.99 [0.90 to 1.00]
  48 weeks | 0.96 [0.87 to 0.99]
  64 weeks | 0.91 [0.81 to 0.96]
  80 weeks | 0.88 [0.78 to 0.94]
  96 weeks | 0.88 [0.78 to 0.94]
  112 weeks | 0.85 [0.74 to 0.92]
  128 weeks | 0.82 [0.71 to 0.89]
  144 weeks | 0.82 [0.71 to 0.89]
  160 weeks | 0.80 [0.69 to 0.88]
  176 weeks | 0.75 [0.63 to 0.84]
  192 weeks | 0.70 [0.57 to 0.80]
  208 weeks | 0.67 [0.54 to 0.77]
  224 weeks | 0.67 [0.54 to 0.77]
  240 weeks | 0.67 [0.54 to 0.77]
  256 weeks | 0.67 [0.54 to 0.77]

ADVERSE EVENTS:
Time Frame: The initial data reported was for the study up to Week 32. This time frame defines the comparative phase of the study where the majority of participants remained on their original randomized assignment and exposure between ruxolitinib and best available therapy was similar. Data inclusive of end of study was reported up to week 256 for Ruxolitinib group. Long term Follow Up for BAT was not reported as all patients have completed the study or crossed over to Ruxolitinib group by week 80.
Description: Safety population: All participants who were enrolled and took at least 1 dose of study medication.
  The initial data reported at Week 32 was based on MedDRA 15.1; the remaining data reported for end of study was based on MedDRA 20.1.
Groups:
- Ruxolitinib - Through Week 32; Ruxolitinib - Week 256 Close Out: Starting dose of 10 mg BID with individualized dose titration ranging from 5 mg QD to 25 mg BID based on safety and efficacy
- Best Available Therapy - Through Week 32: Best Available Therapy (BAT) will be selected by the Investigator for each participant. BAT may not include experimental agents (i.e. those not approved for the treatment of any indication) as well as a limited number of other selected drugs in accordance with the protocol-defined requirements.
Arm/Group | Ruxolitinib - Through Week 32 | Best Available Therapy - Through Week 32 | Ruxolitinib - Week 256 Close Out
Serious Adverse Events (participants affected / at risk) | 15/110 | 10/111 | 44/110
Other Adverse Events (participants affected / at risk) | 105/110 | 104/111 | 107/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib - Through Week 32 (N=110) | Best Available Therapy - Through Week 32 (N=111) | Ruxolitinib - Week 256 Close Out (N=110)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 3
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 1
Glaucoma (Eye disorders) | 1 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 1
Dental necrosis (Gastrointestinal disorders) | 1 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 2
Bronchitis viral (Infections and infestations) | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 5
Vulvovaginitis trichomonal (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Neurological symptom (Nervous system disorders) | 1 | 0 | 1
Bladder disorder (Renal and urinary disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib - Through Week 32 (N=110) | Best Available Therapy - Through Week 32 (N=111) | Ruxolitinib - Week 256 Close Out (N=110)
Anaemia (Blood and lymphatic system disorders) | 20 | 3 | 38
Headache (Nervous system disorders) | 18 | 21 | 25
Diarrhoea (Gastrointestinal disorders) | 16 | 8 | 30
Fatigue (General disorders) | 16 | 17 | 22
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 25 | 30
Dizziness (Nervous system disorders) | 13 | 11 | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 2 | 19
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 5 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 7 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 20
Nasopharyngitis (Infections and infestations) | 10 | 9 | 19
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 12 | 19
Weight increased (Investigations) | 6 | 1 | 26
Abdominal pain (Gastrointestinal disorders) | 10 | 13 | 16
Constipation (Gastrointestinal disorders) | 9 | 3 | 14
Herpes zoster (Infections and infestations) | 7 | 0 | 19
Asthenia (General disorders) | 8 | 12 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 17
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 9 | 13
Nausea (Gastrointestinal disorders) | 7 | 4 | 15
Oedema peripheral (General disorders) | 7 | 7 | 9
Abdominal pain upper (Gastrointestinal disorders) | 6 | 5 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 9
Gamma-glutamyltransferase increased (Investigations) | 6 | 3 | 9
Haematoma (Vascular disorders) | 6 | 3 | 11
Tinnitus (Ear and labyrinth disorders) | 6 | 3 | 9
Insomnia (Psychiatric disorders) | 5 | 6 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 8 | 7
Paraesthesia (Nervous system disorders) | 5 | 7 | 7
Decreased appetite (Metabolism and nutrition disorders) | 3 | 6 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 4
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 7
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 7
Vomiting (Gastrointestinal disorders) | 0 | 0 | 6
Oedema (General disorders) | 0 | 0 | 7
Pyrexia (General disorders) | 0 | 0 | 17
Bronchitis (Infections and infestations) | 0 | 0 | 14
Influenza (Infections and infestations) | 0 | 0 | 13
Pharyngitis (Infections and infestations) | 0 | 0 | 6
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 10
Urinary tract infection (Infections and infestations) | 0 | 0 | 10
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 6
Alanine aminotransferase increased (Investigations) | 0 | 0 | 7
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 7
Blood cholesterol increased (Investigations) | 0 | 0 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 7
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 10
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 16
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 8
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 7
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 6
Neuralgia (Nervous system disorders) | 0 | 0 | 6
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 6
Hypertension (Vascular disorders) | 0 | 0 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.